CLINICAL TRIAL: NCT06814444
Title: Study of the Immunological Infiltrate and Immunometabolic Immunometabolic Profile of Patients with Acute Leukaemia
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: IMMET-2021
Record Dates: First submitted 2024-12-01; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-12

CONDITIONS: Acute Leukemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood (PB) and bone marrow (BM) samples at different time-points, which will be compared with samples obtained from healthy control subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
LThe main aim of this project is to provide an immunophenotypic and immunometabolic characterisation of patients with Acute Leukaemia, before and after therapy, and to understand how changes in the immune system impact the response to therapy.

Specifically:

1. The association between the molecular and metabolic characteristics of leukaemic cells and those of the surrounding immune system will be assessed, in order to identify immune-modulatory metabolic mechanisms activated by malignant cells.
2. The association between immunometabolic signatures and response to therapies will be assessed.
3. The role of EVs as a vehicle for metabolic units capable of regulating the metabolism of immune system cells will be explored.

DETAILED DESCRIPTION:
Multicentre biological study, aimed at collecting and characterising human tissue isolated from acute leukaemia patients. In the context of routine care visits, peripheral blood (PB) and bone marrow (BM) samples will be taken from these patients at different time-points, which will be compared with samples obtained from healthy control subjects.Patients belonging to the haematology OU of the IRCCS AOU of Bologna and to the haematology OUs of the participating centres, suffering from acute leukaemia, will be enrolled. They must be eligible for a treatment scheme that includes either conventional chemotherapy or innovative therapies, such as monoclonal antibodies, molecular therapies with specific targets, metabolic and immunological therapies, as part of the normal care pathway. It is also planned to enrol healthy donors whose samples will be provided by:

* IRCCS AOU of Bologna Immunohaematology and Transfusion Medicine Service (buffy coat)
* Italian Association against Leukaemia, Lymphoma and Myeloma in Bologna (AIL BOLOGNA ODV), within the Haematology Unit of the IRCCS AOU of Bologna (peripheral blood).

ELIGIBILITY:
Inclusion Criteria:

PATIENT

* Diagnosis of Acute Leukaemia.
* Eligibility for a treatment scheme involving either conventional chemotherapy or innovative therapies, such as monoclonal antibodies, molecular therapies with specific targets, metabolic and immunological therapies.
* age ≥ 18 years.
* Signature of informed consent by patients at the time of diagnosis.

Healthy donors (AIL BOLOGNA ODV volunteers)

* age ≥ 18 years.
* Signature of informed consent.

Exclusion Criteria:

* no one

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients belonging to the UOC of Haematology of the IRCCS AOU of Bologna and to the OUs of Haematology OUs of the participating centres, suffering from Acute Leukaemia who, as part of the normal care pathway and completely independently from participation in the study, shall be eligible for a treatment scheme involving either conventional chemotherapy or innovative therapies, such as monoclonal antibodies, molecular therapies with specific targets, therapies metabolic and immunological therapies.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2029-12-11 (Estimated); Study Completion 2030-12-11 (Estimated)

PRIMARY OUTCOMES:
the association between the molecular and metabolic characteristics of leukaemic cells and those of the surrounding immune system, in order to identify immuno-modulatory metabolic mechanisms implemented by malignant cells | Once the sample is collected, through study completion, an average of 1 year
  molecular and metabolic characterisation of the bone marrow infiltrate
the association between immunometabolic signatures and response to therapies | Once the sample is collected, through study completion, an average of 1 year
  evaluation of the immunometabolic profile pre- and post therapy and possible relapse
the role of EVs as a vehicle for metabolic units capable of regulating the metabolism of immune system cells | Once the sample is collected, through study completion, an average of 1 year
  Characterisation of the vesicular component EV and by modulating various metabolic

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Curti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy